CLINICAL TRIAL: NCT06971302
Title: The Effect of Mindfulness Based Breastfeeding Education Given During Pregnancy on Mothers' of Breastfeeding Self-Efficacy Perception, Effectiveness and Mindful
Brief Title: Effect of Mindfulness Based Breastfeeding Education on Mothers' Breastfeeding Parameters
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Ozge Dalgalar, Specialist nurse, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 78017789/050.01.04/2621454
Record Dates: First submitted 2025-04-17; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Breastfeeding
Keywords: minfulness; nursing care; breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: randomize control
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Initially, the pregnant women were administered the Informed Consent Form, the Pregnant Women's Descriptive Characteristics Form, and the Antenatal Breastfeeding Self-Efficacy Scale.No intervention was applied to the pregnant women in the control group. After the first application of the Prenatal Breastfeeding Self-Efficacy Scale, the same scale was applied again six weeks later. Participants were asked to notify the researcher when they gave birth.
  The following instruments were applied to mothers at 1 and 8 weeks postpartum:
  * Postpartum Mother-Baby Identifier Form,
  * Postpartum Breastfeeding Self-Efficacy Scale,
  * Bristol Breastfeeding Assessment Tool, and
  * Mindful Breastfeeding Scale.
  In order to eliminate possible ethical concerns regarding the control group, breastfeeding education was provided to mothers in the control group after the data collection process was completed.
- Mindfulness based breastfeeding education (Experimental): Before the Mindfulness-Based Breastfeeding Education began, the pregnant women were administered the Informed Consent Form, the Pregnant Women's Descriptive Characteristics For.The Mindfulness-Based Breastfeeding Education was delivered to the pregnant women in the intervention group by the researcher both face-to-face and online on the predetermined days and times. The training was supported with visual presentations, videos, and models prepared by the researcher to make it memorable and easy to understand.
  After the final session of the six-week training program, the Antenatal Breastfeeding Self-Efficacy Scale was administered to the participants. The mothers were asked to inform the researcher when they gave birth.
  In the 1st and 8th weeks postpartum, the following forms and scales were administered to the mothers:
  * Postpartum Mother-Infant Descriptive Form,
  * Postnatal Breastfeeding Self-Efficacy Scale,
  * Bristol Breastfeeding Assessment Tool,
  * Mindful Breastfeeding Scale.
  Interventions: Other: Mindfullnes Based Breastfeeding Education

INTERVENTIONS:
Other: Mindfullnes Based Breastfeeding Education — Pregnant women in the intervention group will receive mindfulness-based breastfeeding training, conducted face-to-face and online by the researcher at designated days and times. The intervention group will undergo a total of 12 sessions of mindfulness-based breastfeeding training over a six-week period. The training will be made memorable and easy to understand through the support of visual presentations, videos, and models prepared by the researcher.
  Arms: Mindfulness based breastfeeding education

SUMMARY:
Pregnant women followed at the Tece Family Health Center were contacted via telephone and informed about the study. Pregnant women who expressed interest in participating were assessed according to the inclusion and exclusion criteria using the "Eligibility Assessment Form" prepared by the researcher. Those who met the research criteria were randomly assigned to either the intervention or the control group.

Before starting the Mindfulness-Based Breastfeeding Education, all participants in both groups were asked to complete the Informed Consent Form, the Pregnant Women's Descriptive Characteristics Form, and the Antenatal Breastfeeding Self-Efficacy Scale.

The Mindfulness-Based Breastfeeding Education was delivered to the pregnant women in the intervention group by the researcher, both face-to-face and online, on predetermined days and times. The training was supported with visual presentations, videos, and models prepared by the researcher to make the content more memorable and easier to understand. After the final session of the six-week training program, the participants completed the Antenatal Breastfeeding Self-Efficacy Scale. Mothers were asked to inform the researcher when they gave birth. In the 1st and 8th weeks postpartum, the following were administered: Postpartum Mother-Infant Descriptive Form, Postnatal Breastfeeding Self-Efficacy Scale, Bristol Breastfeeding Assessment Tool, and Mindful Breastfeeding Scale.

No intervention was applied to the pregnant women in the control group. Six weeks after the first administration of the Antenatal Breastfeeding Self-Efficacy Scale, the same scale was administered again. Mothers were asked to notify the researcher when they gave birth. In the 1st and 8th weeks postpartum, the following forms and scales were administered: Postpartum Mother-Infant Descriptive Form, Postnatal Breastfeeding Self-Efficacy Scale, Bristol Breastfeeding Assessment Tool, and Mindful Breastfeeding Scale.

In order to eliminate any potential ethical concerns related to the control group, breastfeeding education was provided to the mothers in the control group after the data collection process had been completed.

DETAILED DESCRIPTION:
The content of the Mindfulness-Based Breastfeeding Education was developed by the researchers based on a comprehensive review of the relevant literature. To evaluate the appropriateness of the educational content, feedback was obtained from expert faculty members with academic experience in breastfeeding and/or mindfulness-related studies.

A list of pregnant women being followed at the Tece Family Health Center was compiled, and those who were interested in participating were provided with general information about the study. Additionally, the researcher shared her contact information with these pregnant women.

Pregnant women who expressed willingness to participate and contacted the researcher were assessed for eligibility using a "Eligibility Assessment Form" prepared by the researcher. Those who met the inclusion criteria were randomly assigned to either the intervention or the control group. The participants were then asked to complete the Informed Consent Form, Pregnant Women's Descriptive Characteristics Form, and the Antenatal Breastfeeding Self-Efficacy Scale.

To facilitate communication with the intervention group, a WhatsApp group was created. Taking into account the needs of the participants and previous studies, appropriate days and times were scheduled for the six-week Mindfulness-Based Breastfeeding Education Program, consisting of weekly two-hour sessions. Participants in the intervention group were divided into subgroups of no more than seven individuals each.

In total, the intervention group received 12 sessions of mindfulness-based breastfeeding education, delivered according to the scheduled days and times. To minimize participant dropout, the program was delivered over six weeks, with the first three weeks conducted online and the remaining three weeks conducted face-to-face, each session lasting two hours.

The educational content covered the following themes: introduction to mindfulness, awareness of the body and the "automatic pilot" mode, mindful communication, coping with difficult emotions and situations, integrating mindfulness into daily life, the postpartum period, and the themes of closure and new beginnings. Mindfulness practices were integrated into the breastfeeding experience under each theme.

No intervention was applied to the control group during the six-week period. At the end of the six weeks, both the intervention and control groups completed the Antenatal Breastfeeding Self-Efficacy Scale once again.

After childbirth, mothers whose newborns did not meet the inclusion criteria were excluded from the sample, and new participants were recruited accordingly. IIn the 1st and 8th weeks postpartum, the Postpartum Mother-Infant Descriptive Form, Postnatal Breastfeeding Self-Efficacy Scale, Bristol Breastfeeding Assessment Tool (BBAT), and the Mindful Breastfeeding Scale (MIND-BFS) were administered to both the intervention and control groups.

To address any potential ethical concerns related to the control group, breastfeeding education was provided to the mothers in the control group following the completion of data collection.

ELIGIBILITY:
Inclusion Criteria:

For pregnant women:

* Who are 18 years or older,
* Who are literate,
* Who are in their 24th to 28th week of pregnancy,
* Who are expecting a singleton pregnancy,
* Who are willing to participate in the study,
* Whose breastfeeding self-efficacy score is below 57,
* Who agree to home visits postpartum for interviews,
* Who do not have any health issues that would prevent breastfeeding,
* Who do not have any communication barriers.

Exclusion Criteria:

For pregnant women who:

* Are under 18 years old,
* Are illiterate,
* Have a gestational age less than 24 weeks or greater than 28 weeks,
* Have a multiple pregnancy,
* Do not wish to breastfeed,
* Have any health issues that would prevent breastfeeding (such as mastectomy, medication use, HIV, etc.),
* Do not speak Turkish,
* Have any psychiatric issues,
* Have a breastfeeding self-efficacy score higher than 57,
* Cannot attend more than two sessions for any reason during the study period,
* Are illiterate,
* Do not sign the Informed Consent Form,
* Do not agree to home visits postpartum for interviews.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 61 (Estimated)
Dates: Start 2024-08-08 (Actual); Primary Completion 2025-03-25 (Actual); Study Completion 2025-08-12 (Estimated)

PRIMARY OUTCOMES:
Breastfeeding evaluated using the Antenatal Breastfeeding Self-Efficacy Scale | during pregnancy, when the study was started and 6 weeks later
  The lowest possible score on the scale is 14, and the highest possible score is 70. There is no cut-off point for the scale, and an increase in the score indicates higher breastfeeding self-efficacy.
Breastfeeding evaluated using the Postnatal Breastfeeding Self-Efficacy Scale | Change from postpartum 1st and 8th week
  The lowest possible score on the scale is 14, and the highest possible score is 70. There is no cut-off point for the scale, and an increase in the score indicates higher Change from breastfeeding self-efficacy.

SECONDARY OUTCOMES:
Breastfeeding evaluated using the Bristol Breastfeeding Assessment Tool | Change from postpartum 1st and 8th week
  The lowest score on the scale is 0, and the highest score is 8. Low scores indicate that breastfeeding is not effective, while high scores indicate that breastfeeding is effective.

OTHER OUTCOMES:
Breastfeeding evaluated using the Mindful Breastfeeding Scale | Change from postpartum 1st and 8th week
  The total score from the scale ranges from 9 to 45, and as the total score increases, the level of awareness in breastfeeding also increases.

CONTACTS AND LOCATIONS:
Overall Officials: DUYGU VEFİKULUÇAY YILMAZ, PROF, Study Chair — Mersin University Faculty of Nursing; ÖZGE DALGALAR, MASTER, Principal Investigator — Mersin University Faculty of Nursing
Locations (1):
- Turkey, Mersin University, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No